CLINICAL TRIAL: NCT02871713
Title: A Randomized Controlled Trial Comparing Intrathecal Morphine with Quadratus Lumborum Block As Part of a Multimodal Analgesia Strategy for Post-cesarean Delivery Analgesia
Brief Title: A Randomized Controlled Trial Comparing Intrathecal Morphine with Quadratus Lumborum Block for Post-cesarean Delivery Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: IWK Health Centre (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Vishal Uppal, Anesthesiologist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1021219
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cesarean Section
Keywords: quadratus lumborum block
MeSH Terms: interventions — Ropivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intrathecal morphine (Active Comparator): Intrathecal morphine 100 mcg
  Interventions: Other: Intrathecal Morphine with 100 mcg morphine
- Quadratus lumborum block (Experimental): Bilateral QLB with 20 ml of 0.5% ropivacaine per side (maximum total dose 3 mg/kg)
  Interventions: Other: Bilateral Quadratus lumborum block with 0.5% ropivacaine
- Intrathecal morphine + Quadratus lumborum block (Experimental): Bilateral QLB with 20 ml of 0.5% ropivacaine per side (maximum total dose 3 mg/kg) + Intrathecal morphine 100 mcg
  Interventions: Other: Bilateral Quadratus lumborum block with 0.5% ropivacaine; Other: Intrathecal Morphine with 100 mcg morphine

INTERVENTIONS:
Other: Bilateral Quadratus lumborum block with 0.5% ropivacaine — Bilateral Quadratus lumborum block with 0.5% ropivacaine
  Arms: Intrathecal morphine + Quadratus lumborum block; Quadratus lumborum block
Other: Intrathecal Morphine with 100 mcg morphine — Intrathecal Morphine with 100 mcg morphine
  Arms: Intrathecal morphine; Intrathecal morphine + Quadratus lumborum block

SUMMARY:
Pain after caesarean delivery (CD) can interfere with the moms' ability to look after her baby and may contribute to developing long term pain and disability. Women having a CD receive pain medication (morphine) as part of their spinal anesthetic to help with pain relief after surgery. Morphine works well however has several side effects such as nausea, vomiting and itching which may be severe enough to make it difficult to care for herself and her new baby. In some cases, morphine causes difficulty in passing urine within first 24-hours of the CD requiring catheterization and thus restricting mobilization. The quadratus lumborum block (QLB) is a newer nerve block that uses local anaesthetic solution to numb the nerves carrying pain sensation from surgical incision site. QLB may be able to provide effective pain control without the side-effects associated with the spinal morphine. This study is to determine if women receiving QLB have as good pain control with fewer side effects than those who do receive the spinal morphine. Adequate pain control will be assessed by their pain scores and recovery in the 24 to 48 hours after CD. The side effect profile of the two techniques, quality of recovery and long term impact will also be compared during this study.

In addition, we would like to compare the patients who received both analgesic regimens (ITM and QLB) with patients who received only one analgesic intervention (i.e. either ITM or QLB). Further, the study will help us answer if combining the two analgesic interventions if beneficial or not.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent CD with planned spinal anesthesia
* American Society of Anesthesia physical status class I & II;
* Age ≥18 years;
* Term gestational age (≥37 weeks);
* Singleton pregnancy;
* English-speaking.

Exclusion Criteria:

* Morbid Obesity (BMI ≥35 kg/m2);
* Subjects with significant obstetric or neonatal co-morbidities;
* Patient enrollment in another study involving medication within 30 days of CD;
* Any other condition, which may impair patients ability to co-operate with data collection;
* Patient height less than 152 cm (5'0");
* History of opioid tolerance or sensitivity;
* Intolerance to non-steroidal anti-inflammatory drugs (NSAIDs);
* Women with a history of illicit drug use or prescribed opioids or benzodiazepines.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Quality of recovery (QoR) score | 24 hours

SECONDARY OUTCOMES:
Morphine equivalent consumption | 24 hours and 48 hours
  morphine equivalent consumption in the 24-h and 48-h period after spinal insertion
Quality of recovery (QoR) score | 48 hours
Incidence of nausea/vomiting needing treatment | 24 hours
Incidence of itching needing treatment. | 24 hours
Incidence of respiratory depression needing treatment. | 24 hours
Worst pain scores | 24 hours
  The primary outcome will be highest pain intensity during first 24-h as measured

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Carvalho B. Respiratory depression after neuraxial opioids in the obstetric setting. Anesth Analg. 2008 Sep;107(3):956-61. doi: 10.1213/ane.0b013e318168b443. PMID 18713913
- [Background] Loane H, Preston R, Douglas MJ, Massey S, Papsdorf M, Tyler J. A randomized controlled trial comparing intrathecal morphine with transversus abdominis plane block for post-cesarean delivery analgesia. Int J Obstet Anesth. 2012 Apr;21(2):112-8. doi: 10.1016/j.ijoa.2012.02.005. Epub 2012 Mar 10. PMID 22410586
- [Background] McKeen DM, George RB, Boyd JC, Allen VM, Pink A. Transversus abdominis plane block does not improve early or late pain outcomes after Cesarean delivery: a randomized controlled trial. Can J Anaesth. 2014 Jul;61(7):631-40. doi: 10.1007/s12630-014-0162-5. Epub 2014 Apr 24. PMID 24764186
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500